CLINICAL TRIAL: NCT03180697
Title: Clinical Study on the Efficacy of Amide Proton Transfer Magnetic Resonance Imaging in Predicting the Efficacy of Bevacizumab in Recurrent Malignant Gliomas
Brief Title: The Efficacy of APT Magnetic Resonance Imaging in Predicting the Efficacy of Bevacizumab in Recurrent Malignant Gliomas
Acronym: APT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: APT MRI and bevacizumab
Record Dates: First submitted 2017-05-11; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Diagnoses Disease; Glioma of Brain
Keywords: Amide Proton Transfer; bevacizumab; recurrent malignant gliomas; efficacy
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen obtained by sugery or biopsy should be retained and test by pathology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- APT MR imaging: Patients who will receive target therapy( Bevacizumab) for recurrent malignant gliomas will be asked to participate in this study. The routine sequences, Gd- enhanced MR imaging and APT MR imaging will be performed before and after target therapy.
  Interventions: Diagnostic Test: APT MR Imaging

INTERVENTIONS:
Diagnostic Test: APT MR Imaging — Patients who will receive target therapy( Bevacizumab) for recurrent malignant gliomas will obtain routine sequences, Gd- enhanced MR imaging and APT MR imaging will be performed before and after target therapy. We will observe the change of tumor after target therapy using APT imaging. We will compare the change of tumor between Gd-enhanced and APT Imaging before and after therapy.

SUMMARY:
Targeted therapy with bevacizumab is the main method to prolong the progression-free survival of patients with recurrent malignant gliomas in recent years. Using noninvasive imaging methods to predict which RMG may respond to bevacizumab regimen therapy is a clinical problem ; on the other hand, repeated gadolinium enhancement may increase the risk of gadolinium ion deposition of brain tissue. Furthermore,there may be a false response phenomenon and cause assessment bias.in the evaluation of treatment efficacy,owing to bevacizumab is only anti-tumor angiogenesis.

Amide Proton Transfer (APT) is a new molecular imaging technique. Our previous studies have shown that imaging features and signal changes of APT can fully reflect the therapeutic effect of malignant glioma,without the injection of contrast agent and avoid the side effects.

RMG patients will be recruited in this study . This project will be designed multi-center, prospective, observational clinical research. The changes of APT signal intensity before and after treatment will be compared with those of different types of RMG line. The relationship between APT imaging characteristics and clinical end point events will be investigated and compared with conventional MR imaging technique. The sensitivity, specificity and accuracy of the progression-free survival and median overall survival will be measured after treatment with bevacizumab.

DETAILED DESCRIPTION:
Recurrent Malignant Gliomas (RMG) have a very short survival time, and re-operation risk is large and failed to significantly improve the prognosis of patients. At present, targeted therapy with bevacizumab is effective in prolonging the progression of patients However, a considerable proportion of recurrent malignant gliomas are insensitive to bevacizumab, and therefore, using noninvasive imaging methods to predict which RMG is sensitive to bevacizumab therapy prior to targeted therapy is very important On the other hand, the current evaluation of bevacizumab is mainly based on the degree of gadolinium enhancement and tumor volume changes, repeated gadolinium injection may increase the risk of gadolinium ion deposition of brain tissue, and because of Bevacizumab only acting as an anti-tumor angiogenesis, and a false response may occur in assessing efficacy, which is a bias in the overall assessment of bevacizumab.

Amide Proton Transfer (APT) is a new molecular imaging technique for the detection indirect of free protein and peptide concentrations based on chemical saturation exchange. Our previous studies have shown that APT signal is independent of gadolinium-enhanced imaging markers , The signal intensity is closely related to the density of tumor cells, cell proliferation and angiogenesis. Therefore, the imaging features and signal changes of APT can fully reflect the therapeutic effect of malignant glioma, and avoid the side effects caused by contrast injection.

This study will be designed as multi-center, prospective, observational clinical research. 100 cases of RMG patients in Zhujiang Hospital and Nanfang Hospital will be recruited. The patients will be examined with conventional MRI and APT-MRI imaging of 3.0T high field MRI. The treatment of different types of RMG line will be scanned with APT protocol. The changes of signal intensity will be studied. The relationship between APT imaging characteristics and clinical end point events will be observed and compared with conventional MR imaging technique. Two techniques will be used to predict the the 6-month progression-free survival after bevacizumab treatment. The aim of this study is to determine whether APT can predict the efficacy of bevacizumab in the treatment of RMG, and which RMG is effective and sensitive to bevacizumab therapy .Also,we will evaluate the feasibility of APT-MR imaging as a surrogate biomarker for predicting the efficacy of targeted therapy and to establish the basic criteria for the selection of individualized targeted therapy regimens for RMG.

ELIGIBILITY:
Inclusion Criteria:

1. malignant glioma patients at least 4 weeks after surgery;
2. after radiotherapy or chemotherapy after the recurrence, stop to put,
3. the age of patients ≥ 18 years old;
4. bone marrow, liver and kidney function is good;
5. not using steroid hormones or disabled for more than 5 days;
6. patients are generally in good condition, expected survival is greater than 8 weeks, Karnofsky test is greater than 60.

Exclusion Criteria:

1. patients with refractory hypertension, active vascular disease, bleeding, intestinal perforation and other medical history;
2. frail and difficult to tolerate treatment;
3. HIV positive;
4. pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with recurrent maligant glioma will be recuritted. All the patients are eligible for the inclusive criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-03 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Signal intensity of tumor on APT imaging | From date of confirmed recurrence until the date of deterioration or date of death from any cause. That means measure, assessed APT signal intensity at 6 weeks, 12 weeks,18 weeks and so on, assessed up to 1 year.
  Observe the change of signal intensity of tumor on APT MR imaging before and after therapy, determine the predictive value of APT imaging about the efficacy of Bevacizumab in recurrent malignant gliomas.

SECONDARY OUTCOMES:
Dimension of tumor on Gd-enhanced MRI | Measure tumor dimension at 6 weeks, 12 weeks and 18 weeks for the most. It will be ended at any time the patient dies.
  Observe the change in dimension of recurrent tumor on Gd-enhanced MRI

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxiao Wu, Master, Principal Investigator — Institutional Ethics Review Board
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No